CLINICAL TRIAL: NCT01496365
Title: A Randomized, Double-Blind, Placebo and Active Comparator-Controlled Study of DS-5565 for Treatment of Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Treatment of Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS5565-A-U201
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Keywords: pain, diabetes, neuropathy
MeSH Terms: conditions — Diabetes Mellitus | interventions — mirogabalin; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- DS-5565 5mg nighttime (Experimental): DS-5565 5 mg/day (one 5 mg tablet at bedtime)
  Interventions: Drug: DS-5565 tablet; Drug: placebo capsule
- DS-5565 10 mg at bedtime (Experimental): DS-5565 10 mg/day (one 10 mg tablet at bedtime)
  Interventions: Drug: DS-5565 tablet; Drug: placebo capsule
- DS-5565 15 mg at bedtime (Experimental): DS-5565 15 mg/day (one 5 mg tablet plus one 10 mg tablet at bedtime)
  Interventions: Drug: DS-5565 tablet; Drug: placebo capsule
- DS-5565 20 mg total per day (Experimental): DS-5565 20 mg/day (one 10 mg tablet in the morning and one 10 mg tablet at bedtime)
  Interventions: Drug: DS-5565 tablet; Drug: placebo capsule
- DS-5565 30 mg total per day (Experimental): DS-5565 30 mg/day (one 5 mg tablet plus one 10 mg tablet in the morning and one 5 mg tablet plus one 10 mg tablet at bedtime)
  Interventions: Drug: DS-5565 tablet; Drug: placebo capsule
- Pregabalin 300 mg total per day (Active Comparator): Pregabalin 300 mg/day (two 150 mg capsules, in the morning and at bedtime)
  Interventions: Drug: pregabalin capsule; Drug: Placebo tablet

INTERVENTIONS:
Drug: DS-5565 tablet — 5mg and 10mg tablets
  Arms: DS-5565 10 mg at bedtime; DS-5565 15 mg at bedtime; DS-5565 20 mg total per day; DS-5565 30 mg total per day; DS-5565 5mg nighttime
Drug: pregabalin capsule — 75mg and 150mg over-encapsulated
  Other Names: Lyrica
  Arms: Pregabalin 300 mg total per day
Drug: Placebo tablet
  Other Names: placebo tablet matching DS-5565 tablet
  Arms: Pregabalin 300 mg total per day
Drug: placebo capsule
  Other Names: placebo capsule matching over-encapsulated pregabalin
  Arms: DS-5565 10 mg at bedtime; DS-5565 15 mg at bedtime; DS-5565 20 mg total per day; DS-5565 30 mg total per day; DS-5565 5mg nighttime

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effectiveness of DS-5565 compared to placebo (inactive substance) and pregabalin in diabetic subjects with DPN.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy (DPN) affects up to 50% of patients who have diabetes for at least 25 years. Up to 26% of all patients with DPN experience neuropathic pain. DPN pain contributes to sleep disorders, depression, and anxiety, which together may have an impact on a patient's well-being and quality of life.

There are currently several drugs used to treat painful DPN. For example, Lyrica® (pregabalin) is approved by the United States Food and Drug Administration (FDA) to treat neuropathic pain associated with DPN and is commonly prescribed. The dosage of the FDA-approved drugs is limited by side-effects such as dizziness, sleepiness, weight gain and swelling of the hands, legs, and feet. As a result, many patients suffering from DPN pain do not get satisfactory pain relief.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years of age
2. Able to give informed consent and willing to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures
3. Type 1 or type 2 diabetes with a hemoglobin A1c (HbA1c) ≤ 10% at Screening and on a stable antidiabetic medication regimen for at least 30 days prior to Screening (insulin therapy is acceptable)
4. Painful distal symmetrical sensorimotor polyneuropathy (as per American Society of Pain Educators guidelines ) diagnosed for at least 6 months, based on neurological history and/or examination; diagnosis includes absent or reduced deep tendon reflexes at both ankles
5. At Screening, a pain score of ≥ 40 mm on the SF-MPQ VAS
6. At Randomization, a pain score of ≥ 40 mm on the SF-MPQ VAS and an ADPS of ≥ 4 on the 11-point NRS, the latter calculated from a minimum of 4 pain ratings in daily diaries obtained during the 1-week Baseline Period (prior to randomization)
7. Creatinine clearance > 60 mL/min (estimated using the Cockcroft-Gault equation)
8. Antidiabetic and other medications anticipated to remain stable and constant during the study period
9. Women of child bearing potential (WOCBP) must be using an adequate method of contraception as detailed in the protocol to avoid pregnancy during the study and for 4 weeks after study completion

Exclusion Criteria:

1. Diagnosis of mononeuropathy
2. Use of concomitant medications that may confound assessments of efficacy and/or safety (see Section 5.2)
3. Major psychiatric disorders
4. Have had a malignancy other than basal cell carcinoma within the past 2 years
5. At Visit 1, have a white blood cell count < 2500/mm3, neutrophil count < 1500/mm3, or platelet count < 100 x 103/mm3
6. Clinically significant unstable diabetes mellitus, unstable hepatic, respiratory, or hematologic illness, unstable cardiovascular disease (including myocardial infarction in the 3 months prior to Visit 1), or symptomatic peripheral vascular disease
7. Clinically significant findings on the Screening ECG
8. History of pernicious anemia, untreated hypothyroidism, chronic hepatitis B, hepatitis B within the past 3 months, or human immunodeficiency virus infection
9. Amputations of body parts other than toes
10. Prior therapeutic failure of pregabalin or gabapentin (considered unresponsive or intolerant to treatment); therapeutic failure implies lack of efficacy following full titration to effective doses (eg, 300 mg/day for pregabalin)
11. Known hypersensitivity to pregabalin or gabapentin
12. Requirement for concomitant anticonvulsant and antidepressant therapy, with the exception of stable doses of SSRIs
13. Neurologic disorders unrelated to DPN that may confound the assessment of pain associated with DPN
14. Skin conditions that could alter sensation
15. Other sources of pain that may confound assessment or self-evaluation of the pain due to DPN
16. Abuse of prescription medications, street drugs or alcohol (including alcohol dependence) within the last 1 year
17. Current enrollment in another investigational study, participation in another investigational study with the past 30 days, or other current or recent use of any investigational drug
18. Pregnancy (as based on lab test results) or breast feeding
19. Laboratory values exceeding limits listed in Table 4.1 of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2012-09-07 (Actual); Study Completion 2012-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Merante, MD, Study Director — Daiichi Sankyo
Locations (69):
- United States (69):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Buena Park, California
  - Burbank, California
  - Chino, California
  - Fresno, California
  - Huntington Beach, California
  - Lakewood, California
  - Lomita, California
  - Long Beach, California
  - Santa Monica, California
  - Walnut Creek, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Golden, Colorado
  - Cromwell, Connecticut
  - Fairfield, Connecticut
  - Bradenton, Florida
  - Brooksville, Florida
  - Clearwater, Florida
  - Hallandale, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Sunrise, Florida
  - Columbus, Georgia
  - Gainesville, Georgia
  - Marietta, Georgia
  - Evansville, Indiana
  - Madisonville, Kentucky
  - Paducah, Kentucky
  - Hyattsville, Maryland
  - Brockton, Massachusetts
  - Farmington Hills, Michigan
  - Olive Branch, Mississippi
  - Florissant, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Albany, New York
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Greensburg, Pennsylvania
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Chattanooga, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Renton, Washington
  - Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 452 participants who met all inclusion criteria and no exclusion criteria were enrolled and randomized in the study at 80 clinic sites in the United States.
Pre-assignment Details: Participants were randomized to 1 of 7 treatment groups which included placebo, pregabalin 150 mg BID, DS-5565 5 mg QD, DS-5565 10 mg QD, DS-5565 15 mg QD, DS-5565 10 mg BID, and DS-5565 15 mg BID.
Groups:
- Placebo: Participants who were randomized to placebo.
- Pregabalin 150 mg BID: Participants who were randomized to pregabalin 150 mg twice daily (BID).
- DS-5565 5mg QD: Participants who were randomized to DS-5565 5 mg every day (QD).
- DS-5565 10 mg QD: Participants who were randomized to DS-5565 10 mg every day (QD).
- DS-5565 15 mg QD: Participants who were randomized to DS-5565 15 mg every day (QD).
- DS-5565 10 mg BID: Participants who were randomized to DS-5565 10 mg twice daily (BID).
- DS-5565 15 mg BID: Participants who were randomized to DS-5565 15 mg twice daily (BID).
Period: Overall Study
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Started | 112 | 56 | 57 | 57 | 57 | 56 | 57
Completed | 97 | 41 | 51 | 53 | 44 | 46 | 51
Not Completed | 15 | 15 | 6 | 4 | 13 | 10 | 6
Not completed — Adverse Event | 2 | 3 | 3 | 2 | 5 | 6 | 4
Not completed — Withdrawal by Subject | 6 | 6 | 0 | 1 | 3 | 2 | 1
Not completed — Protocol Violation | 2 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Other | 4 | 4 | 2 | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline and demographic characteristics are reported in All Enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID | Total
Number analyzed (Participants) | 112 | 56 | 57 | 57 | 57 | 56 | 57 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.57) | 59.5 (9.40) | 58.9 (9.85) | 60.9 (9.92) | 61.4 (8.70) | 60.4 (8.59) | 59.3 (8.54) | 60.1 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 24 | 30 | 28 | 23 | 24 | 25 | 210
  Male | 56 | 32 | 27 | 29 | 34 | 32 | 32 | 242
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 3 | 1 | 0 | 4 | 1 | 1 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 4
  Black or African American | 27 | 17 | 11 | 9 | 12 | 10 | 8 | 94
  White | 81 | 36 | 45 | 43 | 44 | 44 | 46 | 339
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 112 | 56 | 57 | 57 | 57 | 56 | 57 | 452

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 5 in Average Daily Pain Score (ADPS) Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: Average daily pain score (ADPS) is a participant-reported instrument that measures pain intensity using an 11-point numeric rating scale (NRS) where 0 is defined as no pain and 10 is defined as worst possible pain. Higher scores indicate worse pain intensity level. The change from baseline to Week 5 is reported where a negative value is considered an improvement in pain intensity. A minimally meaningful effect was defined as a decrease of at least 1.0 point [scale of 0 to 10] versus placebo).
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: ADPS was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
units on a scale | -1.86 (2.18) | -1.79 (2.27) | -2.04 (2.22) | -2.32 (2.17) | -2.66 (2.37) | -2.64 (2.45) | -2.79 (2.43)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.8916, ANCOVA; Least squares mean = -0.05, 95% CI 2-sided [-0.81 to 0.70]
Statistical Analysis 2: Comparison: Placebo vs DS-5565 5mg QD; Test type: Superiority; p = 0.5569, ANCOVA; Least squares mean = -0.22, 95% CI 2-sided [-0.95 to 0.51]
Statistical Analysis 3: Comparison: Placebo vs DS-5565 10 mg QD; Test type: Superiority; p = 0.1544, ANCOVA; Least squares mean = -0.53, 95% CI 2-sided [-1.25 to 0.20]
Statistical Analysis 4: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0137, ANCOVA; Least squares mean = -0.94, 95% CI 2-sided [-1.69 to -0.19]
Statistical Analysis 5: Comparison: Placebo vs DS-5565 10 mg BID; Test type: Superiority; p = 0.0171, ANCOVA; Least squares mean = -0.88, 95% CI 2-sided [-1.61 to 0.16]
Statistical Analysis 6: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0060, ANCOVA; Least square means = -1.01, 95% CI 2-sided [-1.74 to -0.29]
Statistical Analysis 7: Comparison: Pregabalin 150 mg BID vs DS-5565 5mg QD; Test type: Superiority; p = 0.7051, ANCOVA; Least squares mean = -0.17, 95% CI 2-sided [-1.03 to 0.69]
Statistical Analysis 8: Comparison: Pregabalin 150 mg BID vs DS-5565 10 mg QD; Test type: Superiority; p = 0.2772, ANCOVA; Least squares mean = -0.47, 95% CI 2-sided [-1.33 to 0.38]
Statistical Analysis 9: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0458, ANCOVA; Least squares mean = -0.89, 95% CI 2-sided [-1.77 to -0.02]
Statistical Analysis 10: Comparison: Pregabalin 150 mg BID vs DS-5565 10 mg BID; Test type: Superiority; p = 0.0569, ANCOVA; Least squares mean = -0.83, 95% CI 2-sided [-1.69 to 0.02]
Statistical Analysis 11: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0271, ANCOVA; Least squares mean = -0.96, 95% CI 2-sided [-1.81 to -0.11]

2. Secondary Outcome: Least Square Means of Average Daily Pain Score by Week Mixed Effects Model for Repeated Measures (MMRM) Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: Average daily pain score (ADPS) is a participant-reported instrument that measures pain intensity using an 11-point numeric rating scale (NRS) where 0 is defined as no pain and 10 is defined as worst possible pain. Higher scores indicate worse pain intensity level. The least square means of ADPS (assessed by MMRM) are reported where a negative value is considered an improvement in pain intensity. A minimally meaningful effect was defined as a decrease of at least 1.0 point [scale of 0 to 10] versus placebo).
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: ADPS was assessed in the Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
units on a scale
  Week 1 | -0.55 [-0.81 to -0.29] | -1.10 [-1.49 to -0.72] | -0.68 [-1.04 to -0.31] | -0.95 [-1.31 to -0.58] | -1.13 [-1.51 to -0.75] | -1.26 [-1.62 to -0.89] | -1.40 [-1.76 to -1.04]
  Week 2: number analyzed (Participants) | 106 | 48 | 55 | 54 | 47 | 53 | 57
  Week 2 | -1.12 [-1.47 to -0.77] | -1.75 [-2.26 to -1.24] | -1.38 [-1.86 to -0.89] | -1.56 [-2.04 to -1.07] | -1.76 [-2.28 to -1.25] | -1.72 [-2.20 to -1.23] | -2.33 [-2.80 to -1.85]
  Week 3: number analyzed (Participants) | 102 | 45 | 53 | 54 | 44 | 48 | 55
  Week 3 | -1.47 [-1.86 to -1.08] | -1.79 [-2.36 to -1.21] | -1.62 [-2.17 to -1.08] | -1.78 [-2.32 to -1.23] | -2.30 [-2.88 to -1.72] | -2.38 [-2.93 to -1.82] | -2.55 [-3.08 to -2.02]
  Week 4: number analyzed (Participants) | 100 | 44 | 52 | 53 | 44 | 47 | 52
  Week 4 | -1.67 [-2.08 to -1.26] | -1.83 [-2.45 to -1.22] | -2.01 [-2.59 to -1.44] | -2.41 [-2.98 to -1.83] | -2.46 [-3.08 to -1.85] | -2.68 [-3.27 to -2.10] | -2.72 [-3.29 to -2.15]
  End of treatment: number analyzed (Participants) | 97 | 41 | 51 | 53 | 44 | 46 | 52
  End of treatment | -1.91 [-2.35 to -1.47] | -1.87 [-2.53 to -1.21] | -2.05 [-2.66 to -1.44] | -2.40 [-3.01 to -1.80] | -2.90 [-3.56 to -2.25] | -2.87 [-3.49 to -2.24] | -2.79 [-3.39 to -2.19]

3. Secondary Outcome: Average Daily Pain Score Responder Rates Based on ≥30% and ≥50% Decrease From Baseline at Endpoint) Following Treatment With DS-5565 or Placebo Compared to Pregabalin
Description: Average daily pain score (ADPS) is a participant-reported instrument that measures pain intensity using an 11-point numeric rating scale (NRS) where 0 is defined as no pain and 10 is defined as worst possible pain. Higher scores indicate worse pain intensity level.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: ADPS was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
Participants
  Responder rate: ≥30% decrease from baseline: Yes | 45 | 19 | 22 | 32 | 34 | 34 | 32
  Responder rate: ≥30% decrease from baseline: No | 63 | 31 | 33 | 24 | 17 | 22 | 25
  Responder Rate: ≥50% decrease from baseline: Yes | 26 | 14 | 11 | 16 | 20 | 24 | 25
  Responder Rate: ≥50% decrease from baseline: No | 82 | 36 | 44 | 40 | 31 | 32 | 32

4. Secondary Outcome: Mean Change From Baseline to End-of-Treatment in Average Daily Sleep Interference Score Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: Average Daily Sleep Interference Score (ADSIS) is the weekly average of patient-reported sleep interference (rated every morning on a numerical scale of 0 = "pain did not interfere with sleep" to 10 = "pain completely interfered with sleep" over the past 24 h), where higher scores indicate worse outcome.The change from baseline to Week 5 in ADSIS is being reported as the average of the last 7 available daily scores. The greater the negative value, the greater the improvement in sleep.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: ADSIS was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 50 | 56 | 57
units on a scale | -1.98 (2.38) | -1.94 (2.08) | -2.19 (2.35) | -2.35 (2.31) | -2.97 (2.57) | -2.52 (2.89) | -2.69 (2.43)

5. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ) Sensory and Affective Scores Change From Baseline to Endpoint Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: The SF-MPQ sensory score is the sum of 11 pain descriptors each scored from 0 to 3:
  throbbing, shooting, stabbing, sharp cramping, gnawing, hot-burning, aching, heavy, tender, and splitting. Thus, the SF-MPQ sensory score ranges from 0 to 33, where lower scores indicate a better outcome. The SF-MPQ affective score is the sum of four pain descriptors each scored from 0 to 3: tiring-exhausting, sickening, fearful, and punishing cruel. Thus, SF-MPQ affective score ranges from 0 to 12, where lower scores indicate a better outcome. The change from baseline to Week 5 in SF-MPQ sensory and affective scores are being reported. The greater the negative value, the greater the improvement in sensory and affective scores.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: SF-MPQ sensory and affective scores were assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
units on a scale
  Sensory score: number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 55 | 56
  Sensory score | -6.29 (6.77) | -5.94 (7.32) | -8.02 (6.62) | -8.73 (6.70) | -6.86 (6.77) | -6.56 (7.42) | -8.55 (6.84)
  Affective score: number analyzed (Participants) | 108 | 50 | 55 | 55 | 51 | 55 | 56
  Affective score | -2.10 (2.93) | -1.98 (3.19) | -2.35 (2.80) | -2.44 (3.07) | -1.84 (2.28) | -1.40 (3.19) | -2.23 (2.74)

6. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ) Total Score and Visual Analog Scale Change From Baseline to Endpoint Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: The SF-MPQ sensory score is the sum of 11 pain descriptors each scored from 0 to 3: throbbing, shooting, stabbing, sharp cramping, gnawing, hot-burning, aching, heavy, tender, and splitting. Thus, the SF-MPQ sensory score ranges from 0 to 33, where lower scores indicate a better outcome. The SF-MPQ affective score is the sum of four pain descriptors each scored from 0 to 3: tiring-exhausting, sickening, fearful, and punishing cruel. Thus, SF-MPQ affective score ranges from 0 to 12, where lower scores indicate a better outcome. The SF-MPQ total score comprises the sum of the sensory and affective scores. The SF-MPQ VAS ranges from 0 (no pain) to 100 (worst possible pain), where lower scores indicate a better outcome. The change from baseline to Week 5 in SF-MPQ total score and VAS are being reported. The greater the negative value, the greater the improvement in total score (sensory and affective scores) and VAS pain.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: SF-MPQ total score and VAS pain were assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 55 | 51 | 55 | 56
units on a scale
  Total score | -8.39 (8.91) | -7.92 (9.89) | -10.36 (8.54) | -11.16 (9.29) | -8.71 (8.11) | -7.96 (9.77) | -10.79 (8.94)
  VAS pain | -20.84 (25.12) | -19.28 (24.27) | -27.40 (22.52) | -28.56 (23.67) | -28.73 (26.73) | -25.45 (25.46) | -32.82 (26.97)

7. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ) Present Pain Intensity Change From Baseline to Endpoint Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: The SF-MPQ present pain intensity ranges from 0 (no pain) to 5 (excruciating), where lower scores indicate a better outcome. The change from baseline to Week 5 in SF-MPQ present pain intensity is being reported. The greater the negative value, the greater the improvement in present pain intensity.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: SF-MPQ present pain intensity was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
units on a scale | -0.85 (1.21) | -0.84 (0.96) | -1.00 (0.86) | -1.04 (1.23) | -0.90 (1.03) | -0.73 (1.34) | -1.02 (1.15)

8. Secondary Outcome: Mean Change From Baseline to Endpoint of Modified Brief Pain Inventory (BPI) Subscale, Interference With Daily Functions, Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: The Modified Brief Pain Inventory (BPI) includes Interference with Daily Functions Subscale, Worst Pain Intensity, Least Pain Intensity, Average Pain Intensity, Pain Right Now, and Relief From Pain. The range of interference subscale is 0-10, where lower scores indicate a better outcome. The change from baseline to Week 5 in Modified Brief Pain Inventory is being reported. The greater the negative value, the greater the improvement in interference with daily functions.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: Modified BPI was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
units on a scale | -1.5 (2.11) | -1.7 (1.83) | -1.6 (1.97) | -2.5 (2.11) | -2.4 (2.35) | -2.1 (2.51) | -2.6 (2.34)

9. Secondary Outcome: Mean Change From Baseline to Endpoint of Modified BPI Subscales, Worst, Least and Average Pain Intensity, Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: The Modified Brief Pain Inventory (BPI) includes Interference with Daily Functions Subscale, Worst Pain Intensity, Least Pain Intensity, Average Pain Intensity, Pain Right Now, and Relief From Pain. The range of worst pain intensity in the last 24 hours is 0-10, where lower scores indicate a better outcome. The range of least pain intensity in the last 24 hours is 0-10, where lower scores indicate a better outcome. The range of average pain intensity in the last 24 hours is 0-10, where lower scores indicate a better outcome. The change from baseline to Week 5 in Modified Brief Pain Inventory is being reported. The greater the negative value, the greater the improvement in worst, least, and average pain intensity.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: Modified BPI was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
units on a scale
  Worst Pain Intensity: number analyzed (Participants) | 107 | 50 | 55 | 55 | 51 | 55 | 57
  Worst Pain Intensity | -2.1 (2.53) | -1.9 (2.61) | -2.0 (2.26) | -2.6 (2.53) | -2.7 (2.71) | -2.3 (3.06) | -3.0 (3.09)
  Least Pain Intensity: number analyzed (Participants) | 107 | 50 | 55 | 55 | 51 | 55 | 57
  Least Pain Intensity | -1.3 (2.37) | -0.9 (1.98) | -1.6 (2.55) | -1.7 (2.69) | -2.0 (2.31) | -1.0 (2.58) | -1.9 (2.20)
  Average Pain Intensity: number analyzed (Participants) | 107 | 50 | 55 | 55 | 51 | 55 | 57
  Average Pain Intensity | -1.7 (2.16) | -1.5 (1.95) | -1.7 (2.18) | -2.3 (2.31) | -2.0 (2.34) | -1.8 (2.72) | -2.3 (2.22)

10. Secondary Outcome: Mean Change From Baseline to Endpoint of Modified BPI Subscale, Pain Right Now, Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: The Modified Brief Pain Inventory (BPI) includes Interference with Daily Functions Subscale, Worst Pain Intensity, Least Pain Intensity, Average Pain Intensity, Pain Right Now, and Relief From Pain. The range of pain right now is 0-10, where lower scores indicate a better outcome. The change from baseline to Week 5 in Modified Brief Pain Inventory is being reported. For pain right now, the greater the negative value, the greater the improvement.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: Modified BPI was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
units on a scale | -2.0 (2.35) | -1.8 (1.94) | -2.0 (2.13) | -2.5 (2.44) | -2.5 (2.36) | -2.0 (3.09) | -2.5 (2.75)

11. Secondary Outcome: Mean Change From Baseline to Endpoint of Modified BPI Subscale, Relief From Pain, Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: The Modified Brief Pain Inventory (BPI) includes Interference with Daily Functions Subscale, Worst Pain Intensity, Least Pain Intensity, Average Pain Intensity, Pain Right Now, and Relief From Pain. The range of % relief from pain is 0-100, where higher scores indicate a better outcome. The change from baseline to Week 5 in Modified Brief Pain Inventory is being reported. For relief from pain, the higher the score, the greater the improvement in pain relief.
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: Modified BPI was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
score on a scale | 26.4 (37.67) | 20.4 (31.06) | 31.5 (34.72) | 32.0 (36.33) | 23.0 (37.39) | 35.3 (33.13) | 33.0 (43.52)

12. Secondary Outcome: Patient Global Impression of Change at End-of-Treatment or Early Termination Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: Patient Global Impression of Change (PGIC) has a range of 7 possible responses for overall status since start of the study, where 0 was defined as 'Very much improved' and 7 was defined as 'Very much worse'. Lower scores indicate a better outcome. PGIC was analyzed based on the following definitions: Participant's overall status was minimally improved or better (ie, score ≤3) or Participant's overall status was much improved or better (ie, score ≤ 2).
Time Frame: Baseline up to Week 5 postdose, up to 10 months total follow up
Population: PGIC was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 51 | 56 | 57
Participants
  Overall status is much improved or better (score ≤2): number analyzed (Participants) | 106 | 50 | 55 | 55 | 50 | 52 | 56
  Overall status is much improved or better (score ≤2): Yes | 33 | 19 | 27 | 30 | 24 | 25 | 28
  Overall status is much improved or better (score ≤2): No | 73 | 31 | 28 | 25 | 26 | 27 | 28
  Overall status is minimally improved or better (score ≤3): number analyzed (Participants) | 106 | 50 | 55 | 55 | 50 | 52 | 56
  Overall status is minimally improved or better (score ≤3): Yes | 66 | 33 | 45 | 46 | 37 | 38 | 44
  Overall status is minimally improved or better (score ≤3): No | 40 | 17 | 10 | 9 | 13 | 14 | 12

13. Secondary Outcome: Drug-related Treatment-Emergent Adverse Events (n ≥2 Participants in Any Treatment Group) Following Treatment With DS-5565 Compared to Pregabalin and Placebo
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) which began or worsened in severity after the first administration of study drug. Drug-related TEAEs included AEs that were considered related to the study drug as judged by the Investigator. TEAEs were classified according to MedDRA 14.1.
Time Frame: From the time of signing the informed consent form (ICF) up to 10 months postdose
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
Number analyzed (Participants) | 108 | 50 | 55 | 56 | 53 | 56 | 57
Participants
  Drug-related TEAEs | 31 | 35 | 24 | 21 | 40 | 34 | 37
  Participants with ≥1 drug-related TEAEs | 20 | 14 | 13 | 12 | 17 | 18 | 19
  Nervous System Disorders | 3 | 7 | 4 | 7 | 9 | 14 | 13
  Dizziness | 1 | 1 | 0 | 5 | 5 | 4 | 7
  Somnolence | 1 | 4 | 1 | 1 | 3 | 5 | 4
  Headache | 1 | 0 | 3 | 3 | 0 | 2 | 1
  Balance disorder | 0 | 2 | 0 | 0 | 1 | 3 | 2
  Amnesia | 0 | 0 | 0 | 0 | 0 | 0 | 2
  General Disorders & Administration Site Conditions | 4 | 4 | 2 | 1 | 6 | 4 | 6
  Fatigue | 1 | 2 | 0 | 1 | 2 | 2 | 2
  Oedema peripheral | 0 | 2 | 2 | 0 | 1 | 2 | 1
  Gastrointestinal Disorders | 5 | 2 | 3 | 3 | 5 | 2 | 2
  Nausea | 1 | 0 | 2 | 1 | 1 | 2 | 1
  Constipation | 1 | 0 | 0 | 2 | 1 | 0 | 2
  Dry mouth | 0 | 1 | 1 | 0 | 2 | 0 | 0
  Psychiatric Disorders | 3 | 5 | 2 | 2 | 3 | 1 | 5
  Insomnia | 1 | 1 | 0 | 0 | 2 | 0 | 1
  Investigations | 4 | 2 | 1 | 2 | 3 | 2 | 2
  Weight increased | 1 | 0 | 0 | 1 | 0 | 2 | 1
  Blood creatinine phosphokinase increased | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Eye Disorders | 2 | 1 | 1 | 0 | 2 | 1 | 2
  Vision blurred | 2 | 1 | 1 | 0 | 2 | 0 | 2
  Reproductive System and Breast Disorders | 0 | 0 | 0 | 0 | 2 | 1 | 1
  Erectile dysfunction | 0 | 0 | 0 | 0 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the time of signing the informed consent form (ICF) up to 10 months postdose in the Safety Analysis Set.
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) which began or worsened in severity after the first administration of study drug.
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 5mg QD | DS-5565 10 mg QD | DS-5565 15 mg QD | DS-5565 10 mg BID | DS-5565 15 mg BID
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/50 | 0/55 | 0/56 | 0/53 | 0/56 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/108 | 0/50 | 2/55 | 3/56 | 2/53 | 1/56 | 0/57
Other Adverse Events (participants affected / at risk) | 48/108 | 30/50 | 29/55 | 28/56 | 30/53 | 33/56 | 36/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Pregabalin 150 mg BID (N=50) | DS-5565 5mg QD (N=55) | DS-5565 10 mg QD (N=56) | DS-5565 15 mg QD (N=53) | DS-5565 10 mg BID (N=56) | DS-5565 15 mg BID (N=57)
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Pregabalin 150 mg BID (N=50) | DS-5565 5mg QD (N=55) | DS-5565 10 mg QD (N=56) | DS-5565 15 mg QD (N=53) | DS-5565 10 mg BID (N=56) | DS-5565 15 mg BID (N=57)
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 7 | 6 | 4 | 9
Headache (Nervous system disorders) | 4 | 2 | 6 | 4 | 1 | 5 | 1
Somnolence (Nervous system disorders) | 1 | 4 | 1 | 1 | 3 | 5 | 7
Balance disorder (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 3 | 3
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 5 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 4 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3 | 3 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1 | 3 | 2 | 1 | 1
Oedema peripheral (General disorders) | 1 | 4 | 2 | 4 | 2 | 3 | 2
Fatigue (General disorders) | 2 | 2 | 0 | 2 | 4 | 2 | 2
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 5 | 4 | 2 | 2 | 0 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 2 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 3 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Crying (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness exertional (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Formication (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous stomatitis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0
Gait disturbance (General disorders) | 2 | 1 | 0 | 0 | 2 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Sluggishness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gravitational oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza-like illness (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 3 | 2 | 1 | 2 | 0 | 1 | 1
Blood glucose increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 2 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Positive rombergism (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine renal clearance abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tandem gait test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Plantar fascitiis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Joint lock (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anger (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 2 | 1 | 0 | 2 | 0 | 2
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No